CLINICAL TRIAL: NCT04555577
Title: Phase I Trial of DNA-PK Inhibitor (M3814) in Combination With Radiation and Adjuvant Temozolomide in Newly Diagnosed MGMT Unmethylated Glioblastoma
Brief Title: Peposertib and Radiation Therapy, Followed by Temozolomide for the Treatment of Patients With Newly Diagnosed MGMT Unmethylated Glioblastoma or Gliosarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1035; NCI-2020-04491 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1035 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-10; First posted 2020-09-18 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — peposertib; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage I (Peposertib, Radiation therapy, Temozolomide) (Experimental): CONCURRENT: Patients undergo standard of care radiation therapy daily (Monday-Friday) for 30 fractions. Patients also receive Peposertib PO on each day of radiation therapy and given 1-2 hours before each treatment fraction. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.
  ADJUVANT: Patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Peposertib; Radiation: Radiation Therapy; Drug: Temozolomide
- Stage II (Peposertib, Radiation, Temozolomide, Surgery) (Experimental): CONCURRENT: Patients receive Peposertib and undergo standard of care radiation therapy as in Stage I. Within 1-14 days after the completion of radiation therapy, patients undergo surgical resection.
  ADJUVANT: Patients receive temozolomide as in Stage I.
  Interventions: Drug: Peposertib; Radiation: Radiation Therapy; Procedure: Resection; Drug: Temozolomide

INTERVENTIONS:
Drug: Peposertib — Given PO
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
  Arms: Stage II (Peposertib, Radiation, Temozolomide, Surgery)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I trial investigates the side effects and best dose of Peposertib, and to see how well it works in combination with radiation therapy in treating patients with newly diagnosed MGMT unmethylated glioblastoma or gliosarcoma. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Peposertib may further stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving Peposertib with radiation therapy may work better than radiation therapy alone in treating patients with glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of Peposertib (M3814) in combination with standard of care radiation dose (60 Gy, 2 Gy/fraction over 6 weeks) in patients with newly diagnosed MGMT unmethylated glioblastoma (GBM). (Stage I) II. To determine the ability of M3814 to cross the blood brain barrier and to evaluate their pharmacodynamic properties in resected tissue. (Stage II)

SECONDARY AND EXPLORATORY OBJECTIVES:

I. To evaluate the dose limiting toxicities (DLT). (Stage I) (Secondary Objective) II. To determine the overall response rate (ORR), median progression free survival (mPFS) and median overall survival (mOS) of M3814 in combination with radiation. (Stage I) (Secondary Objective) II. To determine the overall response rate (ORR), median progression free survival (mPFS) and median overall survival (mOS) of M3814 in combination with radiation. (Stage II) (Exploratory Objective)

CORRELATIVE OBJECTIVES:

I. To evaluate pharmacodynamic properties of M3814. II. To assess the alterations in tumor immune microenvironment as a result of deoxyribonucleic acid (DNA)-dependent protein kinase (DNA-PK) inhibition.

OUTLINE: This is a dose-escalation study of Peposertib. Patients are assigned to 1 of 2 stages.

STAGE I (CONCURRENT): Patients undergo standard of care radiation therapy daily (Monday-Friday) for 30 fractions. Patients also receive Peposertib orally (PO) on each day of radiation therapy and given 1-2 hours before each treatment fraction. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.

STAGE I (ADJUVANT): Patients receive temozolomide PO once daily (QD) on days 1-5. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

STAGE II (CONCURRENT): Patients receive Peposertib and undergo standard of care radiation therapy as in Stage I. Within 1-14 days after the completion of radiation therapy, patients undergo surgical resection.

STAGE II (ADJUVANT): Patients receive temozolomide as in Stage I.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Be willing and able to provide written informed consent for the trial. Participants with cognitive impairment will be enrolled. Cognitive function will be assessed by the treating physician or designee through a neurological examination. The formal consent for such participants will be obtained from their legally authorized representative. For cognitively impaired adults who are enrolling in the study by consent of a legally authorized representative, assent of the subject is required for the subjects with the ability to communicate assent. This assent will be documented in subject fs consent note.
* Age 18 years or older
* Histologically confirmed World Health Organization (WHO) grade 4 glioma (GBM) or gliosarcoma, IDH wild-type, per WHO 2021 classification .IDH status is to be determined by IDH1 R132H immunohistochemistry except for patients ≤ age 54 in whom IDH sequencing will be required to detect non-canonical IDH mutations.
* Have KPS of 3 60 or ECOG . 2 according to appendix 5.
* A baseline MRI of brain obtained no more than 14 days prior to study enrollment on a stable or tapering dose of steroids for at least 3 days
* Demonstrate adequate organ function as defined below.
* All screening labs should be performed within 14 days prior to Day 1 of the study.
* Female subjects of childbearing potential should have a negative serum pregnancy test within 14 days of Day 1 of the study.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile.
* All screening labs should be performed within 14 days prior to Day 1 of the study.
* Female subjects of childbearing potential should have a negative serum pregnancy test within 14 days of Day 1 of the study.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile.
* Female subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception during the course of the study.

Newly diagnosed GBM only

* Documentation of MGMT unmethylated GBM per testing at any Clinical Laboratory Improvement Amendment (CLIA) certified laboratory
* Patients must have undergone brain surgery or biopsy and must not have had any further cancer treatments following surgery Recurrent GBM only
* Any number of recurrences
* Presence of enhancing, resectable disease
* Candidate for re-radiation with ability to meet optic nerve and brainstem departmental dose constraints per treating physicians
* 6 mos or more since last radiation
* Has not received re-radiation for GBM in the past except for stereotactic radiosurgery

Exclusion Criteria:

* Has received prior interstitial brachytherapy or implanted chemotherapy.
* Active treatment with the tumor treating filed devices such as Optune during radiation will be excluded. Concurrent use of Optune during the adjuvant temozolomide cycles is allowed.
* Any serious medical condition that interferes with adherence to study procedures.
* Malignancies other than the disease under study within 2 years prior to Day 1 of the study, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score £ 6, and prostate-specific antigen [PSA] £ 10 mg/mL, etc).
* Has known disease in the posterior fossa, gliomatosis cerebri, leptomeningeal disease, extracranial disease. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating physician.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the screening visit.
* Contraindication for undergoing MRIs.
* Inability to comply with study and follow-up procedures.
* Signs or symptoms of serious infection such as surgical wound infection, received IV antibiotics within 2 weeks prior to Day 1 of the study.

oPatients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.

oPatients receiving oral antibiotics for minor infections such as urinary tract infection are eligible.

* Administration of a live, attenuated vaccine within 4 weeks before Day 1 of the study or anticipation that such a live, attenuated vaccine will be required during the study
* Influenza vaccination can be given. Patients must not receive live, attenuated influenza vaccine (e.g., FluMistâ) within 4 weeks prior to Day 1 of the study or at any time during the study and for 5 months after completion of adjuvant TMZ.
* History of long QT syndrome.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of PEPOSERTIB or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* Anticipation of need for a major surgical procedure during the course of the study (excluding patients in Stage II with planed non-urgent neuro-surgical resection)
* Subjects at increased risk for radiation toxicities, such as known active collagen vascular disease (example; scleroderma, Sjogren's disease, etc) or other inherited radiation hypersensitivity syndromes (example; Gorlin syndrome, Fanconi anemia, ataxia-telangiectasia, etc.)
* Active difficulty swallowing, malabsorption or other chronic gastrointestinal disease or conditions (including pancreas deficiency requiring Creon therapy) that may hamper compliance and/or absorption of PEPOSERTIB.
* Patients may not receive concomitant chemotherapy, immunotherapy, or radiotherapy (other than as pertained to GBM as described in section 1.1) while patients are on study.

Newly diagnosed GBM only

* History of MGMT methylated status performed at any CLIA certified laboratory. Recurrent GBM only
* Prior history of scalp / surgical wound infection or wound dehiscence
* Prior exposure to bevacizumab. Patients in stage II C and D (recurrent GBM) may receive bevacizumab as clinically indicated during the adjuvant phase of treatment (physician choice) once 6 weeks has elapsed from the surgery and if there are no wound healing concerns

Medication-Related Exclusion Criteria:

PEPOSERTIB

• Subjects currently receiving or unable to stop using medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP) 3A, CYP2C19, CYP2C9 and / or P-glycoprotein (P-gp) (CYP and / P-gp must stop at least 1 week before treatment with PEPOSERTIB for inhibitors and 3 weeks before treatment with PEPOSERTIB for inducers) or drugs mainly metabolized by CYP3A, CYP2C19, CYP2C9 with a narrow therapeutic index (must stop at least 1 day prior). Please refer to https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers for a list of drugs metabolized by the above mentioned enzymes. In addition concomitant use of H2 blockers of proton pump inhibitors (PPIs) is prohibited. Patients must stop H2 blockers and PPIs 4 days prior to the first treatment. Calcium carbonate use is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Stage I) | Within the first 10 weeks of study treatment
  Will employ the Bayesian optimal interval to find the MTD.
Ability of Peposertib (M3814) to cross the blood brain barrier (Stage II) | At 1, 2, and 4 hours after drug administration on fraction day 1 and at pre-dose and 1, 2, and 4 hours after drug administration on fraction day 10
  Ability of the investigational drug to cross the blood brain barrier will be tested by measuring concentration of the drug within the blood and the resected brain tumor tissue. This will be correlated with biomarkers of deoxyribonucleic acid (DNA) damage in brain tumor tissue, blood, and hair follicle.

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLT) (Stage I) | Within the first 10 weeks of study treatment
  A DLT is defined as a clinically significant adverse event considered at least possibly related to M3814 in combination with radiation during the first 10 weeks of study treatment (4 weeks after completion of radiation and DNA damage response [DDR] inhibitors) for both stage I and stage II patients.
Overall response rate (Stage I) | Up to 3 years
Median progression-free survival (Stage I) | From study enrollment until time of first occurrence of disease progression, relapse, or death due to disease, assessed up to 3 years
Median overall survival (Stage I) | Up to 3 years
Overall response rate (Stage II) | Up to 3 years
Median progression-free survival (Stage II) | From study enrollment until time of first occurrence of disease progression, relapse, or death due to disease, assessed up to 3 years
  Progression-free survival will be evaluated using the Kaplan-Meier product-limit survival curve methodology and will be compared to historical controls. Median progression free survival will be estimated using Kaplan-Meier estimates and associated two-sided 95% confidence intervals.
Median overall survival (Stage II) | Up to 3 years
  Overall survival will be evaluated using the Kaplan-Meier product-limit survival curve methodology and will be compared to historical controls.

OTHER OUTCOMES:
Pharmacodynamic properties of M3814 | Up to 3 years
  Blood and hair follicle will be obtained from stage I & II patients during the screening period, on days 8-12 of concurrent radiation and M3814, and on the last day of radiation and at disease progression. Logistic regression will be used to explore the correlations between response rates and correlative markers. Changes in correlative markers over time will be analyzed by Wilcoxon signed rank tests for pairs of times and linear mixed effects models more generally. Data graphs will be generated to visualize data distributions as well as relationships between variables.
Alterations in tumor immune microenvironment | Up to 3 years
  Will assess the alterations in tumor immune microenvironment as a result of deoxyribonucleic acid-dependent protein kinase inhibition. Logistic regression will be used to explore the correlations between response rates and correlative markers. Changes in correlative markers over time will be analyzed by Wilcoxon signed rank tests for pairs of times and linear mixed effects models more generally. Data graphs will be generated to visualize data distributions as well as relationships between variables.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Majd, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org